CLINICAL TRIAL: NCT05578937
Title: Correlation Between Musculoskeletal Disorders and the Associated Factors of Healthcare Professionals in the Hospital Setting
Brief Title: Musculoskeletal Disorders and the Associated Factors of Healthcare Professionals
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera SS. Antonio e Biagio e Cesare Arrigo di Alessandria (Other)
Responsible Party: Sponsor
Other Study IDs: DISCOFAS
Record Dates: First submitted 2022-10-11; First posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Musculoskeletal Disorders; Psychosocial Problem
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim is to assess the prevalence of musculoskeletal disorders among Italian health professionals by analysing demographic and psychosocial factors. In addition, the impact of the symptoms detected on the quality of life and physical and mental health was analyzed. All health workers on duty in hospital wards for at least 12 months

DETAILED DESCRIPTION:
The online questionnaire sent to the participants was divided into two sections.

The first section concerned the collection of demographic data of the participants (eg age, gender, level of education, work experience, company to which they belong, department, profession, etc.).

The second section concerned the assessment of the prevalence of musculoskeletal disorders, pain, quality of life and assessment of subjective perception of health and assessment of psychosocial factors in the workplace.

ELIGIBILITY:
Inclusion Criteria:

* health personnel who were active in clinical practice during the study period from January to June 2022.
* All health professionals who signed the informed consent
* Health professionals in service in the wards for at least 12 months from the date of sending the questionnaire.

Exclusion Criteria:

Health workers with unsuitability for handling loads

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The population is represented by all the health workers of the inpatient wards (clinics are excluded as the staff inserted may already be unsuitable for handling loads)
Sampling Method: Non-Probability Sample
Enrollment: 291 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
musculoskeletal disorders | 8 months
  prevalence of musculoskeletal disorders

SECONDARY OUTCOMES:
demographic and psychosocial factors | 8 months
  prevalence of factors and correlation with musculoskeletal disorders

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana Bolgeo, PhD, Principal Investigator — Azienda Ospedaliera SS Antonio e Biagio e Cesare Arrigo, Alessandria, Italy, EU
Locations (1):
- Azienda ospedaliera nazionale SS Antonio e Biagio e Cesare Arrigo, Alessandria, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Milhem M, Kalichman L, Ezra D, Alperovitch-Najenson D. Work-related musculoskeletal disorders among physical therapists: A comprehensive narrative review. Int J Occup Med Environ Health. 2016;29(5):735-47. doi: 10.13075/ijomeh.1896.00620. PMID 27518884
- [Background] Anderson SP, Oakman J. Allied Health Professionals and Work-Related Musculoskeletal Disorders: A Systematic Review. Saf Health Work. 2016 Dec;7(4):259-267. doi: 10.1016/j.shaw.2016.04.001. Epub 2016 Apr 28. PMID 27924228
- [Background] Azma K, Hosseini A, Safarian MH, Abedi M. Evaluation of the Relationship Between Musculoskeletal Discomforts and Occupational Stressors Among Nurses. N Am J Med Sci. 2015 Jul;7(7):322-7. doi: 10.4103/1947-2714.161250. PMID 26258080